CLINICAL TRIAL: NCT01779271
Title: Phase 3 Study of Pelubiprofen & Loxoprofen in Patients With Upper Respiratory Tract Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Plb CD 301 Version 3.10
Record Dates: First submitted 2013-01-21; First posted 2013-01-30 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Acute Upper Respiratory Infection; Fever
Keywords: Pelubi; Pelubiprofen; Loxoprofen; Anti-pyretic; Fever
MeSH Terms: conditions — Fever | interventions — pelubiprofen; loxoprofen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pelubiprofen (Experimental)
  Interventions: Drug: Pelubiprofen
- Loxoprofen (Active Comparator)
  Interventions: Drug: Loxoprofen

INTERVENTIONS:
Drug: Pelubiprofen
  Other Names: Pelubiprofen 30 mg
  Arms: Pelubiprofen
Drug: Loxoprofen
  Other Names: Loxoprofen 60mg
  Arms: Loxoprofen

SUMMARY:
Multi-center, Randomized, Double blind, Controlled Parallel-group Comparative Phase 3 Clinical trial to assess the efficacy and safety of Pelubiprofen Compared to Loxoprofen in patients with Acute upper respiratory infection.

ELIGIBILITY:
Inclusion Criteria:

1. Over 15 years old
2. Male and Female
3. Patients with fever over 38.0°C due to cold (acute upper respiratory tract infection)
4. Patients with upper respiratory tract infection outbreak within 2 days and who did not received drug administration
5. Subjects who voluntarily or legal guardian agreed with written consent

Exclusion Criteria:

1. Fever reducer administration Within 4 hours from the screening point
2. Any incidence of febrile crisis from the past six months
3. Patients with Ulcers, gastrointestinal disorders which are confirmed by endoscopy
4. Patients with continuously administrating gastrointestinal disorder related drug
5. Patients with severe blood damage
6. Severe hepatic impairment (ALT, AST value more than 2 times the upper limit of the normal range)
7. With severe renal impairment (serum creatinine value is more than 2 times the upper limit of the normal range)
8. Patients with severe left ventricular dysfunction

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in Body temperature from baseline | 0, 0.5, 1, 1.5, 2, 3, 4, 6 Hour

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, South Korea, Seoul, South Korea

REFERENCES:
- [Derived] Jang AS, Kim SH, Lee SP, Na MJ, Yoo KH, Park CH, Park SY, Choi BW. The Efficacy and Safety of Pelubiprofen in the Treatment of Acute Upper Respiratory Tract Infection: A Multicenter, Randomized, Double-Blind, Non-Inferiority Phase III Clinical Trial Compared to Loxoprofen. J Clin Med. 2025 Feb 21;14(5):1450. doi: 10.3390/jcm14051450. PMID 40094866